CLINICAL TRIAL: NCT03933228
Title: Ultrasound-Guided Combined Interscalene-Cervical Plexus Versus Combined Supraclavicular-Cervical Plexus Block for Surgical Anesthesia in Clavicular Fractures: A Retrospective Observational Study
Brief Title: Analgesia for Clavicular Fracture and Surgery
Status: Completed | Type: Observational
Sponsor: Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019CZTCWM4
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Clavicular Fractures
Keywords: Combined Interscalene-Cervical Plexus Block; Combined Supraclavicular-Cervical Plexus Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interscalene-Cervical Plexus Block: Ultrasound-Guided Combined Interscalene-Cervical Plexus Block
  Interventions: Procedure: Interscalene-Cervical Plexus Block
- Supraclavicular-Cervical Plexus Block: Ultrasound-Guided Combined Supraclavicular-Cervical Plexus Block
  Interventions: Procedure: Supraclavicular-Cervical Plexus Block

INTERVENTIONS:
Procedure: Interscalene-Cervical Plexus Block — Ultrasound-Guided Combined Interscalene-Cervical Plexus Block
  Groups: Interscalene-Cervical Plexus Block
Procedure: Supraclavicular-Cervical Plexus Block — Ultrasound-Guided Combined Supraclavicular-Cervical Plexus Block
  Groups: Supraclavicular-Cervical Plexus Block

SUMMARY:
Compared efficacy of ultrasound-guided combined interscalene-cervical plexus versus combined supraclavicular-cervical plexus block for surgical anesthesia in clavicular fractures.

DETAILED DESCRIPTION:
The primary objective of this study was to compare the effectiveness of ultrasound-guided combined interscalene-cervical plexus versus combined supraclavicular-cervical plexus block for surgical anesthesia in clavicular fractures.The hypothesis of this study was that the supraclavicular-cervical plexus block could provide better anesthesia with less anesthesia related complications.

ELIGIBILITY:
Inclusion Criteria:

* Surgery of the clavicular fractures under combined cervical plexus plus brachial plexus block
* Urgent or planned surgery

Exclusion Criteria:

* Refused to sign informed consent
* Pregnant women
* Allergic to the local anesthetic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Block success rate | At time 15 minutes after the block
  Sensory blockade was assessed using the pinprick test at the surgery site

SECONDARY OUTCOMES:
Acute complications | At the end of surgery immediately
  Number of participants with phrenic nerve palsy

CONTACTS AND LOCATIONS:
Overall Officials: Ruizhao Lv, M.D, Principal Investigator — Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei, China